CLINICAL TRIAL: NCT02622451
Title: Differential Sensitivity Markers in Youth Drug Abuse Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Natalis Counseling Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1504S69041; R34DA037888 (NIH)
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Adolescent Substance Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Youth Behavioral Intervention (Other): Teen Intervene
  Interventions: Behavioral: Teen Intervene
- Parent Education (Other): Everyday Parenting
  Interventions: Behavioral: Everyday Parenting

INTERVENTIONS:
Behavioral: Teen Intervene — Teen Intervene (TI) is an early intervention program for 12-19 year olds who display early stages of alcohol or drug use. TI uses motivational interviewing, goal setting, and skill training to foster the internal development of responsible decision-making with the goal of choosing attitudes and behaviors that are healthier alternatives to drug use behaviors.
  Arms: Youth Behavioral Intervention
Behavioral: Everyday Parenting — Everyday Parenting is a family-focused intervention that works with parents to provide environmental scaffolding necessary to help teens gradually internalize decision-making skills that reinforce and promote healthy lifestyle alternatives.
  Arms: Parent Education

SUMMARY:
This pilot study conducts feasibility and exploratory intervention outcome research that will lead to the development of a personalized intervention framework that seeks to preempt the progression from early drug use to more chronic abuse and dependency. The study will explore moderators representing two frameworks, risk severity and differential sensitivity. Moderators will be explored in their ability to influence the differential efficacy of two adolescent drug abuse interventions.

DETAILED DESCRIPTION:
This R34 pilot study proposes to conduct feasibility and exploratory intervention outcome research that will lead to the development of a personalized intervention framework for early stage adolescent drug users. The study will explore putative moderators representing two theoretically distinct frameworks and determine whether they are suitable candidates for a subsequent R01 study. One moderation framework is based on risk severity (RS) as reflected by individual differences in delay discounting (DD), a form of impulsive decision making that is positively associated with escalation to more serious levels of abuse and addiction. A second more exploratory framework is based on differential sensitivity (DS) theory. The DS framework stipulates that individuals, due to specific sensitivity factors, vary in their responsiveness to environmental influence such as the influence provided by an intervention. The study will explore DS markers associated with the reward motivational system, including dopaminergic genes, the post-auricular physiological reflex and a high sensory-processing sensitivity trait. An agency-university partnership will collaborate in providing services to 120 adolescents (ages 12-17) who were referred to a community counseling center because of a recent alcohol and/or marijuana incident. Recruitment will select mild/moderate drug users. Participants will be randomized to one of two evidence-based drug abuse interventions. The two interventions offer the same delivery dosage but differ in terms of their mechanism of therapeutic change (i.e., degree of environmental influence). The Teen Intervene program (TI; Winters & Leitten, 2007) is a youth-focused intervention that uses motivational interviewing, goal setting, and skills training to foster the internal development of responsible decision-making with the goal of choosing attitudes and behaviors that are healthier alternatives to drug use behaviors. The Everyday Parenting program (EP; Dishion et al., 2003; 2010) is a family focused-intervention that works with parents to provide environmental scaffolding necessary to help teens gradually internalize decision-making skills that reinforce and promote healthy lifestyle alternatives to drug use. The aims of this R34 are to (1) assess feasibility of recruiting, assessing, and following-up enrolled youth in an intervention trial, (2) assess the ability of staff to implement TI and EP with fidelity, and (3) obtain promising data on moderator and outcome variables that will help answer the question of "what intervention works best for which youth" in a subsequent R01 study.

ELIGIBILITY:
Inclusion Criteria:

* Youth ages 12-17
* Substance Use referral to community partner agency
* Adolescent report of weekly-monthly use of one or more substances within the prior 6 months

Exclusion Criteria:

* Current DSM-5 diagnosis of a severe substance use disorder (i.e. substance dependence)
* Adolescent report of daily use of substance within prior 6 months
* Current or past history of psychosis (including suicidal ideation)
* Pervasive developmental disabilities

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-03-08 (Actual)

PRIMARY OUTCOMES:
Delayed Discounting Task | 4 months post-intervention
  Youth Computer Task
Iowa Gambling Task | 4 months post-intervention
  Youth Computer Task
Urinalysis | 4 months post-intervention
  Adolescents will provide urine samples for urinalysis to test for recent drug usage.
Peer Substance Use Test | 4 months post-intervention
  Youth Report
Peer Delinquency Scale | 4 months post-intervention
  Youth Report
Project Towards No Drug Abuse Survey | 4 months post-intervention
  Youth Report
Alcohol Expectancy Questionnaire | 4 months post-intervention
  Youth Report
Single-item self-efficacy Scale | 4 months post-intervention
  Youth Report
Client Satisfaction Questionnaire | 4 months post-intervention
  Parent & Youth Report
Highly Sensitive Person Scale | 4 months post-intervention
  Parent & Youth Report
Parental Monitoring Instrument | 4 months post-intervention
  Parent & Youth Report
Parenting Relationship Questionnaire (PRQ) | 4 months post-intervention
  Parent Report
Family Problem Solving Communication Index | 4 months post-intervention
  Parent Report
Parental Locus of Control Questionnaire | 4 months post-intervention
  Parent Report
Family Assessment Measure - III | 4 months post-intervention
  Parent Report on family functioning .
Conflict Behavior Questionnaire | 4 months post-intervention
  Parent Report

CONTACTS AND LOCATIONS:
Overall Officials: Gerald August, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- Center for Personalized Prevention Research in Children's Mental Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No